CLINICAL TRIAL: NCT00565565
Title: Proof of Concept Study to Investigate Safety, Tolerability, Pharmacokinetics and the Impact on Pulmonary and Systemic Hemodynamics of a Single Oral Dose of BAY60-4552 in Patients With Biventricular Chronic Heart Failure and Pulmonary Hypertension in a Non-randomized, Non-blinded, Dose Escalation Design.
Brief Title: Single Dose Escalation Study in Patients With Chronic Heart Failure
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12356; 2007-003216-54 (EudraCT Number)
Record Dates: First submitted 2007-10-31; First posted 2007-11-30 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Heart Failure
Keywords: Biventriular chronic heart failure, Pulmonary hypertension
MeSH Terms: conditions — Heart Failure; Hypertension, Pulmonary | interventions — BAY 60-4552

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- BAY60-4552, 1 mg (Experimental): Subjects were planned to receive 1 mg of BAY60-4552 as solution
  Interventions: Drug: BAY60-4552
- BAY60-4552, 2.5 mg (Experimental): Subjects were planned to receive 2.5 mg of BAY60-4552 as tablet
  Interventions: Drug: BAY60-4552
- BAY60-4552, 5 mg (Experimental): Subjects were planned to receive 5.0 mg of BAY60-4552 as tablet
  Interventions: Drug: BAY60-4552
- BAY60-4552, 7.5 mg (Experimental): Subjects were planned to receive 7.5 mg of BAY60-4552 as tablet
  Interventions: Drug: BAY60-4552
- BAY60-4552, 10 mg (Experimental): Subjects were planned to receive 10 mg of BAY60-4552 as tablet
  Interventions: Drug: BAY60-4552

INTERVENTIONS:
Drug: BAY60-4552 — Single dose escalation planned at dose of 1 mg, 2.5 mg, 5 mg, 7.5 mg, and 10 mg

SUMMARY:
This study is to demonstrate the safety and tolerability of a single oral dose of BAY60-4552 in a single dose escalation design. Furthermore, this study examines the changes in hemodynamics after application of the test substance.42 hospitalized stable patients with chronic heart failure will be included. Several measurements will be performed to test how good the drug works and wether there are any unwanted reactions to the drug (e.g. blood tests, ECG, heart rate, blood pressure, adverse events). After a observation period the patient will be discharged from the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic heart failure, undergoing routine invasive measurement of hemodynamic parameters

Exclusion Criteria:

* Acute heart failure or acute decompensated heart failure, need for acute cardiologic intervention or surgery, severe renal or hepatic insufficiency, severe valvular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2007-10; Primary Completion 2008-12 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Change in pulmonary capillary wedge pressure | Pre-dose and up to 6 hr post-dose
Change in mean pulmonary artery pressure | Pre-dose and up to 6 hr post-dose
AUC | Pre-dose and up to 72 hr post-dose
  Area under the plasma concentration vs time curve from zero to infinity after single dose
AUC/D | Pre-dose and up to 72 hr post-dose
  AUC divided by dose (mg)
Cmax | Pre-dose and up to 72 hr post-dose
  Maximum drug concentration in plasma after single dose administration
Cmax/D | Pre-dose and up to 72 hr post-dose
  Cmax divided by dose (mg)
Number of participants with adverse events | Approximately 2 weeks

SECONDARY OUTCOMES:
Mean right atrial pressure | Pre-dose and up to 6 hr post-dose
Systolic pulmonary artery pressure | Pre-dose and up to 6 hr post-dose
Diastolic pulmonary artery pressure | Pre-dose and up to 6 hr post-dose
Heart rate | At pre-study visit, pre-dose and up to 24 hr post-dose
Cardiac output | Pre-dose and up to 6 hr post-dose
Pulmonary vascular resistance | Pre-dose and up to 6 hr post-dose
Pulmonary vascular resistance index | Pre-dose and up to 6 hr post-dose
Systemic vascular resistance | Pre-dose and up to 6 hr post-dose
Systemic vascular resistance index | Pre-dose and up to 6 hr post-dose
Cardiac index | Pre-dose and up to 6 hr post-dose
Mean arterial pressure | Pre-dose and up to 6 hr post-dose
Systemic blood pressure | At pre-study visit, pre-dose and up to 24 hr post-dose
Diastolic blood pressure | At pre-study visit, pre-dose and up to 24 hr post-dose
Dyspnea Score | Pre-dose and up to 48 hr post-dose
  Subject is asked unpersuasively about his/her well-being in comparison to the baseline condition, measured on a 7-point Likert scale.
AUC(0-6) | Pre-dose and up to 6 hr post-dose
  AUC from time 0 to 6 h after study drug intake
AUCnorm | Pre-dose and up to 72 hr post-dose
  AUC divided by dose (mg) per kg body weight
AUC(0-tn) | Pre-dose and up to 72 hr post-dose
  AUC from time 0 to the last data point
AUC(0-tn)norm | Pre-dose and up to 72 hr post-dose
  AUC(0-tn) divided by dose (mg) per kg body weight
Cmax,norm | Pre-dose and up to 72 hr post-dose
  Cmax divided by dose (mg) per kg body weight
tmax | Pre-dose and up to 72 hr post-dose
  Time to reach maximum drug concentration in plasma after single dose
t½ | Pre-dose and up to 72 hr post-dose
  Half-life associated with the terminal slope
Mean residence time | Pre-dose and up to 72 hr post-dose
Total body clearance of drug from plasma calculated after oral administration (apparent oral clearance) | Pre-dose and up to 72 hr post-dose
Apparent volume of distribution associated with the terminal phase (after oral administration) | Pre-dose and up to 72 hr post-dose
Amount of drug excreted via urine | Pre-dose and up to 6 hr post-dose
Percent amount of drug excreted via urine | Pre-dose and up to 6 hr post-dose
Renal clearance of drug | Pre-dose and up to 6 hr post-dose
Renin activity | Pre-dose and up to 24 hr post-dose
Change from baseline of noradrenaline after drug administration | Pre-dose and up to 24 hr post-dose
N-terminal pro-atrial natriuretic peptide | Pre-dose and up to 24 hr post-dose
NT-pro B-type natriuretic peptide | Pre-dose and up to 24 hr post-dose
Big endothelin-1 | Pre-dose and up to 24 hr post-dose
Cystatin C | Pre-dose and up to 24 hr post-dose
Change from baseline of osteopontin after drug administration | Pre-dose and up to 24 hr post-dose
Cyclic guanosine mono-phosphate | Pre-dose and up to 24 hr post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (2):
- Germany (2):
  - Bad Nauheim, Hesse
  - Giessen, Hesse

REFERENCES:
- [Result] Acute hemodynamic response to single oral doses of BAY 60-4552, a soluble guanylate cyclase stimulator, in patients with biventricular heart failure. V Mitrovic, B Swidnicki, A Ghofrani, W Mück, N Kirschbaum, J Mittendorf, J-P Stasch, G Wensing, R Frey, S Lentini. BMC Pharmacology 2009; 9(Suppl 1): P51.
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/